CLINICAL TRIAL: NCT06842550
Title: MAintAin Activity in Arthritis: A Feasibility Study
Acronym: MAintAin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-242; HRCI-HRB-2022-010 (Other Grant/Funding Number: HRB HCRI Arthritis Ireland)
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Arthritis
Keywords: Arthritis; Physical Activity Maintenance; Feasibility; Health coaching
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Maintenance Intervention (Experimental): This is a one armed, non controlled study. Participants will receive up to five health coaching sessions led by a trained provider. The aim is to motivate people to meet their physical activity goals, look at their options, make choices and plans, identify challenges, and help them through these changes related to their physical activity and maintenance. Session 1: One to one session with a physical activity coach Session 2-5: Group sessions with approx. 8-10 other people living with arthritis. In the sessions participants will: • Set, reflect and adapt your activity goals • Learn to problem solve • Develop action plans to build new habits. • Learn about opportunities such as walking groups, aqua aerobics and yoga classes are available in your community • Have the support of peers in the group. Please note that these sessions are not exercise classes.
  Interventions: Behavioral: MAintAin Activity with Arthritis

INTERVENTIONS:
Behavioral: MAintAin Activity with Arthritis — Participants will receive up to five health coaching sessions led by a trained provider. The aim is to motivate people to meet their physical activity goals, look at their options, make choices and plans, identify challenges, and help them through these changes related to their physical activity and maintenance. Session 1: One to one session with a physical activity coach Session 2-5: Group sessions with approx. 8-10 other people living with arthritis. In the sessions participants will: • Set, reflect and adapt your activity goals • Learn to problem solve • Develop action plans to build new habits. • Learn about opportunities such as walking groups, aqua aerobics and yoga classes are available in your community • Have the support of peers in the group. Please note that these sessions are not exercise classes.

SUMMARY:
Best practice guidelines across the world always recommend those living with arthritis to be physically active. Research shows that being active can help people living with arthritis to do the things that they want to do for longer, reduce pain, improve quality of life and protect against getting other health conditions such as heart disease, lung disease and cancer. Whilst various exercise programmes support people with arthritis to be active most individuals reduce their level of PA after completion of a prescribed programme. Staying active in the longer-term is more difficult and there is often a decrease in activity over time. Research has shown that exercise programmes helping people to become active, such as exercise classes, may not always have the right approach and focus during the programme to help people to stay active long-term. It is important to understand if people with arthritis can be supported to maintain their activity levels well in to the future. The investigators have already spoken to people living with arthritis, people involved in arthritis care and those involved in promoting physical activity. The research team brought their feedback and the scientific literature together and shaped a new intervention that suits the needs of people with arthritis and helps them to continue to be physically active. The investiagtors will now ask people living with arthritis to try out the new intervention.

Participants will receive up to five coaching sessions that aim to support people with arthritis to maintain their PA after exiting a structured exercise programme. Sessions will be delivered within community venues in a group setting by a trained provider. Sessions will last approximately between 60 and 90 minutes and will be delivered over a period of approximately 4-months.

Participants may receive a smartwatch with an inbuilt step counter such as Fitbit and diary to record their daily steps or physical activity minutes. The diary will also be used to record physical activity maintenance goals, complete action plans and self-monitor progress to build new habits. Participants can continue to use their own smartwatch if they have one.

The research team are interested to know if the programme has any effect on the amount of activity people do over time as well as looking at factors which can help with the understanding of 'why' or 'why not' a PA intervention may have worked.

ELIGIBILITY:
Inclusion Criteria: Those who have exited from a supervised group-based exercise programme for arthritis.

-

Exclusion Criteria: Those aged under 18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview | pre (week zero) and post (week 17)
  Interviews with participants and providers to explore their needs and expectations (pre) and how/if they were met (post)

SECONDARY OUTCOMES:
Physical Activity | pre (week 0) and post (week 17)
  Physical activity data from an accelerometer
Relapse Self Efficacy Questionnaire | pre (week 0) and post (week 17)
  To measure how confident a person is about restarting physical activity
Maintenance Self Efficacy Questionnaire | pre (week 0) and post (week 17)
  To measure how confident a person is about staying physical activity
Self-Report Behavioural Automaticity Index | pre (week 0) and post (week 17)
  To measure physical activity automaticity
Physical Activity Behaviour Self-Evaluation Questionnaire | pre (week 0) and post (week 17)
  To measure opportunity in relation to physical activity
Adapted Action and Coping Planning Questionnaire | pre (week 0) and post (week 17)
  To measure intentions and plans around physical activity
PHYSICAL ACTIVITY REGULATIONS QUESTIONNAIRE (BREQ-3) | pre (week 0) and post (week 17)
  To measure why someone participates why they engage in physical activity
Satisfaction with intervention | post (week 17)
  To measure satisfaction with intervention, using bespoke satisfaction questions and scale (1-5, where 1 is "very dissastified" and 5 is "very satisfied")

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: MAintAin Activity in Arthritis: A study protocol of the co-development and feasibility testing of a physical activity maintenance intervention — https://hrbopenresearch.org/articles/7-75/v1